CLINICAL TRIAL: NCT03920683
Title: Association Between Toe-brachial Index and Coronary Calcification in Asymptomatic Patients with Type 1 and Type 2 Diabetes Mellitus
Brief Title: Toe-brachial Index and Coronary Calcification in Type 1 and 2 Diabetes
Acronym: ACCoDiab
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180409; 2018-A02748-47 (Other: ANSM)
Record Dates: First submitted 2019-01-25; First posted 2019-04-19 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Calcification
Keywords: Prediction of coronary artery calcification score; Diabetes mellitus; Toe-brachial index
MeSH Terms: conditions — Diabetes Mellitus | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diabete type 1 and 2: Data collection from patients treated in the diabetes department, in Pitié-Salpêtrière hospital, and adressed for a one-day hospitalization to assess cardiovascular comorbidities.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Retrospective : data from medical record Prospective : vital statuts from follow-up phone call

SUMMARY:
Diabetes is not a coronary risk equivalent, despite cardiovascular disease is the most common cause of death in diabetes. So, to identify diabetic patients at high cardiovascular risk is necessary. Coronary artery calcification score predicts major coronary events, and improves risk reclassification in asymptomatic diabetic patients. But, cornary artery calcification score is expensive and exposes patients to radiation. So, it cannot be used for large-scale screening. It could be interesting to identify the predictive factors of coronary artery calcification score.

Toe-brachial index is relevant in diabetic patients for the screening of peripheral arterial disease, and predicts cardiovascular events.

The aim of this study is to evaluate the association between toe-brachial index and coronary artery calcification score in asymptomatic patients with type 1 or 2 diabetes. The hypothesis is that toe-brachial index is associated with high coronary artery calcification score. It could be performed first to identify patients who require a coronary artery calcification score. It measurement is reliable, fully automated, repoducible ans cost-effectiveness.

This is a cross-sectional study, with restrospective data collection. All patients addressed to a one-day hospitalization to assess cardiovascular comorbidities are eligible.

Data are collected in patients'medical records. Clinical, biological and imaging data were collected previously during their one-day hospitalization

DETAILED DESCRIPTION:
Cardiovascular disease is the most common cause of death in diabetes. Actually, systematic screening of asymptomatic diabetic patients for silent myocardial ischemia is highly controversial, and is recommended for selected high-risk patients.

Calcium artery calcification score predicts major coronary events, and improves risk reclassification in asymptomatic diabetic patients. The guidelines of the european society of cardiology published in 2013 recommend a screening for silent myocardial ischemia in patients with a high coronary score, without defining a cut-off value. But, assessing cardiovascular risk with calcium coronary score in all asymptomatic patients with diabetes is not feasible. In fact, calcium coronary score expose patients to radiation, is expensive, and is not easily available in health centres. It cannot be used to screen the 4 millions of diabetic patients in France. It could be interesting to identify the predictive factors of a high calcium coronary score, in order to perform coronary artery calcification score only in selected high-risk patients.

Ankle-brachial index is also a marker of cardiovascular risk. Several prospective studies revealed that a low ankle-brachial index predicts cardiovascular events and mortality, and all-cause mortality in diabetes. Nevertheless, a study involving 1343 patients with type 2 diabetes from MESA and Heinz Nixdorf Recall studies has showed that coronary artery calcification score provides better risk reclassification than ankle-brachial index.

Toe-brachial index is particularly relevant in diabetes for peripheral arterial disease screening.

The aim of this study is to evaluate the association between toe-brachial index and coronary artery calcification score in asymptomatic patients with type 1 and 2 diabetes.

The hypothesis is that toe-brachial index is associated with a high coronary artery calcification score. It could be performed first to identify patients who require a coronary artery calcification score. The measurement of toe-brachial index is fully automated, is reliable and reproducible and is cost-effectiveness. This technique is suitable for large-scale screening.

Secondary objectives are :

1. To assess the association between toe-brachial index and severe coronary artery calcification, and to determinate its performance in predicting severe coronary artery calcification
2. To assess the association between toe-brachial index and moderate coronary artery calcification, and to determinate its performance in predicting moderate coronary artery calcification
3. To assess the association between toe-brachial index and the absence of coronary artery calcification, and to determinate its performance in predicting the absence of coronary artery calcification
4. To assess the association between toe-brachial index and early coronary plaque, and to determinate its performance in predicting early coronary atheroma
5. To compare coronary artery calcification between patients with type 1 and type diabetes
6. To assess the association between toe-brachial index and coronary artery calcification in patients with type 1 diabetes
7. To assess the association between toe-brachial index and coronary artery calcification in patients with type 2 diabetes
8. To assess the association between toe-brachial index and an abnormal stress myocardial perfusion tomography, and to determinate its performance in predicting an abnormal stress myocardial perfusion tomography
9. To assess the association between toe-brachial index and an abnormal coronary angiography, and to determinate its performance in predicting an abnormal coronary angiography
10. To assess the association between coronary artery calcification score and an abnormal stress myocardial perfusion tomography, and to determinate its performance in predicting an abnormal stress myocardial perfusion tomography
11. To assess the association between coronary artery calcification score and an abnormal coronary angiography, and to determinate its performance in predicting an abnormal coronary angiography

This is a cross-sectional and single-centre study, with retrospective data collection. All patients addressed to a one-day hospitalization to assess cardiovascular comorbidities, between January 2014 and May 2017, in the diabetes department, in the Pitié-Salpêtrière hospital in Paris, are eligible.

Data are collected in patients' medical records. Clinical, biological and imaging data were collected previously during their one-day hospitalization.

Clinical data are age, sex, diabetes duration, type of diabetes, high blood pressure, dyslipidemia, smoking status, diabetes comorbidities and current medication. Physical examination data are weight, height, body mass index, blood pressure, orthostatic hypotension, symptoms of diabetic peripheral neuropathy, monofilament test, VibraTip and peripheral pulses.

Biological data are HbA1c, fasting blood glucose, HDL-cholesterol, LDL-cholesterol calculated using Friedewald equation, total cholesterol, triglycerides, estimated glomerular filtration rate (eGFR) by modification of diet in renal disease (MDRD), urinary albumin/creatinine ratio, ASAT, ALAT, fibromax protein C reactive and ferritin. Blood and urinary samples have been collected during the one-day hospitalization, and have been analyzed in biochemical department, in Pitié-Salpêtrière hospital.

A retinography bas been performed in patient with known retinopathy or with a mild nonproliferative retinopathy, without ophthalmologic examination since 1 year. Severe retinopathy is defined by severe nonproliferative retinopathy or proliferative retinopathy or retinopathy treated with laser.

Diabetic nephropathy is known or is defined by a urinary albumin/creatinine ratio up to 3 mg/mmol associated with a diabetic retinopathy or a peripheral neuropathy. Albuminuria stages are defined by the urinary albumin/creatinine ratio : no albuminuria if ratio is <3mg/mmol, microalbuminuria if ratio is ≥3 mg/mmol and <30mg/mmol and macroalbuminuria if ratio is ≥30 mg/mmol. Diabetic peripheral neuropathy is known or is defined by typical symptoms or abnormal monofilament test or abnormal ViBratip. Autonomic neuropathy is defined by gastroparesis, cardiovascular autonomic neuropathy, orthostatic hypotension, urinary autonomic dysfunction neuropathy and Charcot foot. Peripheral artery disease is known or is defined by a toe-brachial index <0.7 associated with 2 abnormal pulses on the same side or by a leg artery stenosis ≥ 70% on the ultrasound examination.

Carotid arteries have been studied using an echo-doppler. Intima-media thickness has been measured on longitudinal images, over a 1 cm plaque-free segment free of plaque, 1 cm proximal to the carotid artery bifurcation. Two measurement methods have been used to evaluate intima-media thickness: an automated method using a 3 to 8 MHz linear array transducer (Philips IE33, Koninklijke Philips N.V., Netherlands) and Philips Q-Lab version 8 software (Koninklijke Philips N.V., Netherlands), and a manual method using a 8 or a 4 to 9 MHz transducer (Acuson Sequoi ou Siemens Acuson, respectively). Endpoints are the highest intima-media thickness value between right and left side, and the mean intima-media thickness from right and left side. Plaque is defined as a stenosis <50%, using NASCET and ECST criteria. Carotid stenosis is defined by a stenosis ≥ 50%, using NASCET and ECST criteria.

Toe-brachial index measurement is described in "primary outcome measures". Coronary artery calcification score, stress myocardial perfusion tomography and coronary angiography are described in "secondary outcome measures". Stress myocardial perfusion tomography has been performed if coronary artery calcification score was >100. Coronary angiography has been performed if stress myocardial perfusion tomography was abnormal.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* Diabetes mellitus (type 1 or 2)
* Patients addressed to a one-day hospitalization to assess cardiovascular comorbidities, between January 2014 and May 2017, in the diabetes department, in the Pitié-Salpêtrière hospital
* Coronary artery calcium score available
* Toe-brachial index available

Exclusion Criteria:

* History of coronary artery disease
* History of Raynaud's syndrome
* Opposition of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the diabetes department, in Pitié-Salpêtrière hospital, and adressed for a one-day hospitalization to assess cardiovascular comorbidities.
Sampling Method: Probability Sample
Enrollment: 707 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Toe-brachial index | During the one-day hospitalization in the diabetes department
  Toe-brachial index has been performed by a clinician nurse of the diabetology department, using a fully automatic photoplethysmographic device, Systoe®. Three measurements have been performed on the first toe of both foot : the first one to permit blood volumeflow, and the mean of the others has been recorded to define toe blood pressure. Toe-brachial index is the ratio of toe systolic blood pressure and brachial systolic blood pressure. The lowest value of toe-brachial index between the right and the left side is used. Toe-brachial index cut-off is 0.7.

SECONDARY OUTCOMES:
Vital statuts | Through study completion, an average of 8 months.
  Vital statuts will be collected by the investigator during a follow-up phone call.
Coronary artery calcification | Through study completion, an average of 8 months.
  Coronary artery calcification score has been measured using a cardiac-gated multidetector computerized tomography (semi-automated software using the calcium score developed by Agatston. It is defined as a lesion with a density above 130 Hounsfield units, and with an area above 1mm². Coronary artery calcification score was the amount of the score of left main artery, left anterior descending artery, left circumflex artery and right coronary artery. Standardized categories are used to describe coronary artery calcification score : 0 for absence of calcified plaque, 1 to 10 for minimal plaque, 11 to 100 for mild plaque, 101 to 400 for moderate plaque, and >400 for severe plaque. Age, sex and race-specific percentiles of coronary artery calcification score are also performed, using the methodology described in the Multi-Ethnic Study of Atherosclerosis (validated only for patients between 45 and 84 years old). A score ≥75th percentile defines a high cardiovascular risk.
Stress myocardial perfusion tomography | Through study completion, an average of 8 months.
  Stress myocardial perfusion tomography was realized using a cycloergometer until maximal heart rate (stopped in case of clinical symptoms or ECG abnormalities). Abnormal stress myocardial perfusion tomography is defined by a perfusion defect on stress images on at least one of the 17 anatomical region of the left ventricle, and absent on rest images.
Coronary angiography | Through study completion, an average of 8 months.
  Coronary angiography has been performed in the cardiology department, in Pitié-Salpêtrière hospital. A coronary stenosis is defined by a stenosis≥ 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BOURRON, MD, PhD, Principal Investigator — Assistance Publique Hoptiaux de Paris
Locations (1):
- Diabetology department, Pitié-Salpêtrière hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denimal D, Ponnaiah M, Jeannin AC, Phan F, Hartemann A, Boussouar S, Charpentier E, Redheuil A, Foufelle F, Bourron O. Non-alcoholic fatty liver disease biomarkers estimate cardiovascular risk based on coronary artery calcium score in type 2 diabetes: a cross-sectional study with two independent cohorts. Cardiovasc Diabetol. 2024 Feb 13;23(1):69. doi: 10.1186/s12933-024-02161-x. PMID 38351039